CLINICAL TRIAL: NCT00431444
Title: A Multi-center, Randomized, Double-blind, Double-dummy Study in Postmenopausal Women With Low Bone Mineral Density to Compare the Effects of a Single Dose of i.v. Zoledronic Acid 5 mg, With Daily Oral Raloxifene 60 mg OD on Bone Turnover Markers
Brief Title: Effects of Zoledronic Acid and Raloxifene on Bone Turnover Markers in Postmenopausal Women With Low Bone Mineral Density
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CZOL446HUS121
Record Dates: First submitted 2007-02-01; First posted 2007-02-05 (Estimated); Results first posted 2011-03-11 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-03

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Post-menopausal; Bone mineral density
MeSH Terms: conditions — Osteoporosis | interventions — Raloxifene Hydrochloride; Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Zoledronic Acid (Active Comparator): Zoledronic acid 5 mg (single i.v. infusion) + daily oral placebo for 6 months (zoledronic acid group)
  Interventions: Drug: Zoledronic acid; Drug: Placebo oral pills
- Raloxifene (Active Comparator): Placebo (single i.v. infusion) + oral raloxifene 60 mg/day for 6 months (raloxifene group)
  Interventions: Drug: Raloxifene; Drug: Placebo intravenous (i.v.) infusion

INTERVENTIONS:
Drug: Raloxifene
  Arms: Raloxifene
Drug: Zoledronic acid
  Other Names: Reclast, Aclasta
  Arms: Zoledronic Acid
Drug: Placebo oral pills
  Arms: Zoledronic Acid
Drug: Placebo intravenous (i.v.) infusion
  Arms: Raloxifene

SUMMARY:
This study will compare the effects of Zoledronic acid and Raloxifene in reducing bone turnover markers in postmenopausal women with low bone mineral density over 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Females, between 45 and 80 years (inclusive) of age, considered post-menopausal according to one of the following guidelines:
* Cessation of menses for 18 months in women < 50 years of age
* Cessation of menses for 12 months in women age 50 years or over
* Documented bilateral oophorectomy at least 1 year previously
* Documented T score of less than or equal to -1.5 on dual energy X-ray absorptiometry (DXA) scan at the lumbar spine, total hip or femoral neck within 24 months prior to screening, and clinically indicated for treatment with bisphosphonates (BPs) for osteopenia or osteoporosis
* Signed informed consent prior to initiation of any study procedure

Exclusion Criteria:

* Prior treatment with i.v. bisphosphonates within the last 2 years
* Previous use of oral bisphosphonates within the past 2 years (unless used for less than 8 weeks*).
* *NOTE: If used less than 8 weeks, the washout period is 6 months.
* Treatment with raloxifene, calcitonin, tibolone or hormone replacement therapy. The washout period for these medications is 6 months prior to randomization.
* Any treatment with strontium renalate, sodium fluoride or parathyroid hormone
* Use of systemic high dose corticosteroids at an average dose of ≥ 7.5 mg per day of oral prednisone or equivalent for a period of three months or more within the previous year
* Treatment with any investigational drug within 30 days prior to randomization
* Any woman of child bearing potential
* Patients with fractures occurring within three months prior to randomization
* History of hypersensitivity to bisphosphonates
* History of non-traumatic uveitis or iritis, within 2 years prior to study entry.
* A history of invasive malignancy of any organ system, treated or untreated, within the past 12 months prior to screening; excluding, basal cell or squamous cell carcinoma of the skin, colonic polyps with non-invasive malignancy which have been removed, Ductal Carcinoma in-situ (DCIS) that has been surgically removed, and Carcinoma in-situ (CIS) of the uterine cervix that has been surgically removed.
* Previous major solid organ transplant recipient or on a transplant waiting list
* History of hyperparathyroidism, hypoparathyroidism, Osteogenesis imperfecta, Paget's disease or any metabolic bone disease other than osteoporosis
* Any medical condition which would interfere with the action of the study drug or limit life expectancy to less than 6 months
* Any medical or psychiatric condition which, in the opinion of the investigator, would preclude the participant from adhering to the protocol or completing the trial
* Active dental infection, unhealed dental extraction or planned oral surgery within 3 month prior to randomization.
* Calculated creatinine clearance < 30 mL/min
* Greater than 2+ protein on urine dipstick without evidence of contamination or bacteriuria (may be repeated one time, at least a day apart).
* Serum calcium > 2.75 mmol/L (11.0 mg/dL) or < 2.08 mmol/L (8.3 mg/dL) at screening
* AST, ALT or serum alkaline phosphatase greater than twice the upper limit of normal

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2007-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (17):
- United States (17):
  - Women's Health Research, Phoenix, Arizona
  - Associated Pharma Research Center, Buena Park, California
  - Washington D.C., District of Columbia
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Women's Physicians of Jacksonville, Jacksonville, Florida
  - Tampa Clinical Research, Tampa, Florida
  - Springfield Clinic, Springfield, Illinois
  - Consultants in Women's Health Care, St Louis, Missouri
  - Alegent Health, Omaha, Nebraska
  - Specialty Medical and Research Center, Pahrump, Nevada
  - UMDNJ-Robert Wood Johnson Medical Center, New Brunswick, New Jersey
  - Columbia University, New York, New York
  - Kernodle Clinic, Inc., Burlington, North Carolina
  - The Portland Clinic, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Texas Institute for Clinical Research, Fort Worth, Texas
  - Valley Women's Health Clinic, Renton, Washington

REFERENCES:
- [Derived] Bachmann G, Kriegman A, Goncalves J, Kianifard F, Warren M, Simon JA. Effect of zoledronic acid compared with raloxifene on bone turnover markers in postmenopausal women with low bone density. Menopause. 2011 Aug;18(8):851-6. doi: 10.1097/gme.0b013e31820b80f1. PMID 21796066

RESULTS

PARTICIPANT FLOW:
Groups:
- Zoledronic Acid: Zoledronic acid 5 mg (single intravenous (i.v.) infusion) + daily oral placebo for 6 months (zoledronic acid group)
Period: Overall Study
Arm/Group | Zoledronic Acid | Raloxifene
Started | 56 | 53 (Initially 110 randomized, 1 participant of "Raloxifene" group never took study drug.)
Completed | 51 | 46
Not Completed | 5 | 7
Not completed — Protocol Violation | 1 | 4
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Administrative Problems | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid | Raloxifene | Total
Number analyzed (Participants) | 56 | 53 | 109
Age Continuous [Mean (Standard Deviation); unit: years] | 58.8 (6.97) | 61.5 (8.20) | 60.1 (7.68)
Age, Customized [Number; unit: participants]
  Between 45 and 65 years | 43 | 35 | 78
  >=65 years | 13 | 18 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 53 | 109
  Male | 0 | 0 | 0
Post-menopausal [Mean (Standard Deviation); unit: year] — Number of years the patient had been post-menopausal.
  year | 12.5 (8.94) | 13.4 (9.17) | 13.0 (9.03)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Urine N-telopeptide of Type 1 Collagen (NTx.)
Description: The primary efficacy variable was the change from baseline in urine NTx (corrected by creatinine). The primary analysis time point was at 6 months of treatment. The results are reported as nanomoles (nM) of bone collagen equivalents (BCE) per millimole (mM) of urine creatinine.
Time Frame: Baseline and 6 months
Population: The intent-to-treat (ITT) population consisted of all randomized patients who received at least one dose of study drug and had at least one post-baseline assessment of the primary efficacy variable of urine N-telopeptide of Type 1 collagen (NTx).Observed cases were used, no imputation was performed.
Measure: Mean (Standard Deviation); unit: nM BCE/mM Cr
Arm/Group | Zoledronic Acid | Raloxifene
Number analyzed (Participants) | 52 | 53
nM BCE/mM Cr
  Baseline (n = 52, 53) | 49.054 (20.4515) | 44.460 (23.2789)
  6 months (n = 49, 47) | 23.676 (11.9152) | 34.183 (16.4667)
  Change from baseline to Month 6 (n= 48, 47) | -24.646 (13.9893) | -8.362 (15.3852)

2. Secondary Outcome: Change From Baseline in Urine NTx at 2 Months
Description: The results are reported as nanomoles (nM) of bone collagen equivalents (BCE) per millimole (mM) of urine creatinine.
Time Frame: Baseline and 2 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nM BCE/mM Cr
Arm/Group | Zoledronic Acid | Raloxifene
Number analyzed (Participants) | 54 | 53
nM BCE/mM Cr
  Baseline (n= 52, 53) | 49.054 (20.4515) | 44.460 (23.2789)
  At Month 2 (n= 54, 50) | 17.774 (9.1107) | 40.756 (23.3700)
  Change from baseline to Month 2 (n= 52, 50) | -31.065 (16.4960) | -4.000 (11.2757)

3. Secondary Outcome: Change From Baseline in Urine NTx at 4 Months
Description: The results are reported as nanomoles (nM) of bone collagen equivalents (BCE) per millimole (mM) of urine creatinine.
Time Frame: Baseline and 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nM BCE/mM Cr
Arm/Group | Zoledronic Acid | Raloxifene
Number analyzed (Participants) | 52 | 53
nM BCE/mM Cr
  Baseline (n= 52 , 53) | 49.054 (20.4515) | 44.460 (23.2789)
  At Month 4 (n= 48, 46) | 20.802 (13.1632) | 38.143 (24.9307)
  Change from baseline to Month 4 (n= 47, 46) | -27.832 (15.4142) | -3.920 (17.1348)

4. Secondary Outcome: Change From Baseline in Serum Bone Specific Alkaline Phosphatase (BSAP) at 2 Months
Time Frame: Baseline and 2 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Zoledronic Acid | Raloxifene
Number analyzed (Participants) | 51 | 51
U/L
  Baseline (n= 50, 48) | 30.104 (10.8868) | 27.094 (9.4039)
  At Month 2 (n= 51, 51) | 20.855 (5.8499) | 26.424 (7.8699)
  Change from baseline to Month 2 (n= 47, 46) | -8.947 (6.4181) | -1.085 (4.0969)

5. Secondary Outcome: Change From Baseline in Serum Bone Specific Alkaline Phosphatase (BSAP) at 4 Months
Time Frame: Baseline and 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Zoledronic Acid | Raloxifene
Number analyzed (Participants) | 50 | 48
U/L
  Baseline (n= 50, 48) | 30.104 (10.8868) | 27.094 (9.4039)
  At Month 4 (n= 49, 47) | 18.218 (5.1846) | 25.111 (8.4530)
  Change from baseline to Month 4 (n= 45, 42) | -11.442 (7.8097) | -2.000 (5.0356)

6. Secondary Outcome: Change From Baseline in Serum Bone Specific Alkaline Phosphatase (BSAP) at 6 Months
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Zoledronic Acid | Raloxifene
Number analyzed (Participants) | 51 | 48
U/L
  Baseline (n= 50, 48) | 30.104 (10.8868) | 27.094 (9.4039)
  At Month 6 (n= 51, 47) | 19.237 (5.5181) | 24.981 (7.9932)
  Change from baseline to Month 6 (n= 47, 42) | -10.572 (7.3263) | -2.250 (7.1307)

7. Secondary Outcome: Overall Principal Investigator Satisfaction Assessed by Satisfaction Questionnaire
Description: The investigator was asked to complete satisfaction questionnaires at baseline (Visit 2/Day 1) when each patient's i.v. drug administration occurred. The questionnaire assessed overall satisfaction with the i.v. infusion procedure. The possible answers to the question were: "not at all," "a little," "somewhat," "quite," or "completely."
Time Frame: Immediately after infusion procedure
Population: Intention-to-treat (ITT) population.
Measure: Number; unit: Participants
Arm/Group | Zoledronic Acid | Raloxifene
Number analyzed (Participants) | 54 | 53
Participants
  Not at all / A little | 0 | 0
  Somewhat | 3 | 1
  Quite | 2 | 3
  Completely | 16 | 11
  Missing | 33 | 38

8. Secondary Outcome: Overall Nurse Satisfaction Assessed by Satisfaction Questionnaire
Description: The study coordinator (nurse) was asked to complete satisfaction questionnaires at baseline (Visit 2/Day 1) when each patient's i.v. drug administration occurred. The questionnaire assessed overall satisfaction with the i.v. infusion procedure. The possible answers to the question were: "not at all," "a little," "somewhat," "quite," or "completely."
Time Frame: Immediately after infusion procedure
Population: Intention-to-treat (ITT) population.
Measure: Number; unit: Participants
Arm/Group | Zoledronic Acid | Raloxifene
Number analyzed (Participants) | 54 | 53
Participants
  Not at all / A little / Somewhat | 0 | 0
  Quite | 4 | 3
  Completely | 29 | 35
  Missing | 21 | 15

9. Secondary Outcome: Overall Patient Satisfaction Assessed by Satisfaction Questionnaire
Description: Patients were asked to complete the satisfaction questionnaire at baseline. The questionnaire assessed overall satisfaction with the i.v. infusion procedure. The possible answers to the question were: "not at all," "a little," "somewhat," "quite," or "completely."
Time Frame: Immediately after infusion procedure
Population: Intention-to-treat (ITT) population.
Measure: Number; unit: Participants
Arm/Group | Zoledronic Acid | Raloxifene
Number analyzed (Participants) | 54 | 53
Participants
  Not at all | 1 | 1
  A little | 0 | 1
  Somewhat | 1 | 1
  Quite | 9 | 7
  Completely | 43 | 42
  Missing | 0 | 1

10. Secondary Outcome: Patient Preference at 6 Months for Annual i.v Therapy or Daily Oral Regimens
Description: At the end-of-study visit, Month 6, patients were asked to complete a questionnaire to assess preference for the different treatment modalities (annual i.v. infusion vs. daily oral capsule). The possible answers to question were: "once a year i.v. infusion," "once daily pill," or "both are equal."
Time Frame: At 6 month visit
Population: Intention-to-treat (ITT) population.
Measure: Number; unit: Participants
Arm/Group | Zoledronic Acid | Raloxifene
Number analyzed (Participants) | 54 | 53
Participants
  Once a year intravenous infusion | 47 | 46
  Once daily pill | 3 | 4
  Both are equal | 3 | 3
  Missing | 1 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: The safety population included all randomized patients who received at least one dose of study drug.
Arm/Group | Zoledronic Acid | Raloxifene
Serious Adverse Events (participants affected / at risk) | 1/56 | 1/53
Other Adverse Events (participants affected / at risk) | 31/56 | 13/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid (N=56) | Raloxifene (N=53)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid (N=56) | Raloxifene (N=53)
Constipation (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 5 | 1
Nausea (Gastrointestinal disorders) | 7 | 1
Chills (General disorders) | 3 | 1
Fatigue (General disorders) | 3 | 1
Influenza like illness (General disorders) | 3 | 0
Pain (General disorders) | 4 | 0
Pyrexia (General disorders) | 6 | 0
Sinusitis (Infections and infestations) | 4 | 4
Urinary tract infection (Infections and infestations) | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 3
Headache (Nervous system disorders) | 3 | 0
Hypertension (Vascular disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.